CLINICAL TRIAL: NCT04610645
Title: Live Laser Microscopic Evaluation (OCT) of Radiation Induced Preclinical Alterations of the Skin in Head and Neck Cancer Patients
Brief Title: Optical Coherence Tomography in Patients With Radiotherapy for Head and Neck Cancer
Acronym: ROOCT
Status: Completed | Type: Observational
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Collaborators: Verein zur Forschungsförderung der Krebshilfe OÖ (Unknown); RECENDT GmbH (Unknown); Johannes Kepler Universität Linz, Abteilung FLLL (Unknown); Universitätsklinikum Erlangen (Unknown); Andreas Fahl Medizintechnik-Vertrieb GmbH (Unknown)
Responsible Party: Principal Investigator, Hans Geinitz, Prim. Univ.-Prof. Dr., Krankenhaus Barmherzige Schwestern Linz
Other Study IDs: EKS 39/18
Record Dates: First submitted 2020-10-29; First posted 2020-10-30 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Radiotherapy
Keywords: Optical coherence tomography; OCT; Head and neck cancer; radiotherapy; radiation therapy; skin toxicity; radiation sensitivity; FISH; Quality of Life; EORTC QLQ C30; EORTC H&N 43; Radiochemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — In Situ Hybridization, Fluorescence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Head and Neck Cancer Patients: Patients with adjuvant or definitve radiotherapy or radio-chemotherapy for head and neck cancer
  Interventions: Device: OCT; Device: Dermatoscope; Genetic: 3-Colour FISH

INTERVENTIONS:
Device: OCT — 3x3 OCT volume scans on treated and opposite side of the irreadiated area on head and neck
  Other Names: Lumedica OQlabscope 2.0
Device: Dermatoscope — 2x2 pictures taken with a dermatoscope
  Other Names: Heine iC1 Set/6
Genetic: 3-Colour FISH — Blood sample is examined for breaks per metaphase to determine radiation sensibility of the individual
  Other Names: Fluorescent In Situ Hybridisation

SUMMARY:
The purpose of this study is to determine whether any eventual skin damage caused by radiation therapy can be detected and monitored at a subclinical level via optical coherence tomography (OCT). Another key question is whether subclinical OCT detected skin damage correlates with acute and late clinical toxicity.

DETAILED DESCRIPTION:
Head and neck cancer patients that meet the eligibility criteria and singned the informed consent will undergo OCT-measurements before, during and after the course of radiation therapy. At the same time-points the skin areas are evaluated with dermatoscopy and patients are asked to self-assess their quality of life (EORTC QLQ C30 and respective head and neck module H&N 43). Before the onset of radiation therapy radiation sensitivity analysis will be performed with in-vitro irradion of peripheral blood lymphocytes (FISH).

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer located at: nasopharynx, oropharynx, hypopharynx, larynx, oral cavity and definitive or adjuvant radiation- or radio-chemotherapy

Exclusion Criteria:

* reduced mental capacity
* treatment with C225 Cetuximab
* bearded patients
* overt skin disease
* vast tattoos in the neck region

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutively treated patients with head and neck cancer at the department of radiation therapy Ordensklinikum Linz Barmherzige Schwestern
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
early radiation induced skin structure changes detected in OCT | First week of radiation therapy
  any reproducible difference in skin OCT appearance as compared with baseline (pre-RT)

SECONDARY OUTCOMES:
detection of any skin strucure changes with OCT during the course of RT | weeks 1 - 6 of radiation therapy
  any reproducible difference in skin OCT appearance as compared with baseline (pre-RT)
Correlation of OCT changes with clinical appearent acute side effetcs | weeks 1 - 6 of radiation therapy
  Correlation of OCT changes with CTC radiation toxicity
Correlation of OCT changes with clinical appearent late side effetcs | 1 year post-RT
  Correlation of OCT changes with CTC radiation toxicity
Correlation of OCT changes with radiation sensitivity | OCT: weeks 1-6 of radiation therapy; FISH: pre-RT
  Correlation of OCT with chromosome-breaks per metaphasis in in-vitro irradiated blood lymphocytes (FISH)
Correlation of OCT changes with dermatoscopic skin appearance | weeks 1-6 of RT
  Correlation of OCT changes with standardised evaluated skin appearence via dermatoscopy
Correlation of quality of live with OCT and radiation sensitivity | weeks 1-6 of RT, 6 weeks and 1 year post-RT
  Correlation of quality of live as measured with the EORT QLC C30 and Head and neck module H&N 43 with OCT and radiation sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Hans Geinitz, Prim. Univ.-Prof. Dr., Principal Investigator — Ordensklinikum Linz GmbH Barmherzige Schwestern (Dept. Radiooncology)
Locations (1):
- Department of Radiooncology, Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided